CLINICAL TRIAL: NCT00903240
Title: Phase 3 Study of Bladder Cancer Recurrence Surveillance
Brief Title: Observational Study of Subjects Having Routine Recurrence Screening for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Predictive Biosciences (Industry)
Responsible Party: Ellen Sheets, Predictive Biosciences
Other Study IDs: PBS-001
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2009-11

CONDITIONS: Bladder Cancer Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The specimens to be retained are urine only
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to detect recurrent bladder cancer using a combination of protein and DNA biomarkers in urine

ELIGIBILITY:
Inclusion Criteria:

* Intact bladder
* Scheduled for cystoscopy for transitional cell bladder cancer recurrence screening
* Urine donated prior to cystoscopy, Bladder biopsy, chemotherapy, intravesical therapy, radiation or TUR
* Must be willing to sign IRB approved informed consent

Exclusion Criteria:

* History or current diagnosis of any cancer except transitional cell bladder cancer or basal cell cancer
* Known diagnosis of any autoimmune disease or HIV, HCV or HBV
* History or current TB or any other active infection
* Subject has gross hematuria
* Receiving chemotherapy, intravesical therapy or radiation within 30 days of enrollment
* Any surgery except urologic within past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be from urology and oncology practices
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Sheets, MD, Study Director — Predictive Biosciences
Locations (20):
- United States (20):
  - BCG Oncology, Phoenix, Arizona
  - Urology Associates, Engelwood, Colorado
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Winter Park Urology, Orlando, Florida
  - Metropolitan Urology, Jeffersonville, Indiana
  - Mayo Validation Support Services, Rochester, Minnesota
  - Metro Urology, Woodbury, Minnesota
  - Associates in Urology/Urology Group of NJ, 741 Northfield Avenue, New Jersey
  - Coastal Urology Associates, Brick, New Jersey
  - Capital Regional Urological Surgeons, Albany, New York
  - Community Care Physicians, Albany, New York
  - University Urology Associates, New York, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Associated Medical Professionals, Syracuse, New York
  - The Urology Group, Cincinnati, Ohio
  - Urological Associates of Lancaster, Lancaster, Pennsylvania
  - Triangle Urologic Group, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas